CLINICAL TRIAL: NCT03717311
Title: Pilot Study of the Metabolic Signature of 13C-enriched Wheat Bran Linked to Intestinal Fermentation in Humans: Identification of New Biomarkers
Brief Title: BRAN Pilot Study: Metabolic Signature of Wheat Bran Related to Gut Fermentation in Humans
Acronym: FITABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0143
Record Dates: First submitted 2018-07-11; First posted 2018-10-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: biomarkers; fermentation; labeled wheat bran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 13C enriched bran biscuit (Experimental): The volunteers will consume 5 biscuits (100g) enriched with 13C bran with a 200 ml hot beverage in 15 minutes
  Interventions: Other: Nutritional Intervention

INTERVENTIONS:
Other: Nutritional Intervention — The intervention will be done on 1 day, time during which, each subject will stay at the CRNH. A breakfast containing the fibers will be given to them, then during 24h a following will be done to get fecal, urinary, plasmatic and expiratory samples. Standardized lunch, dinner and collation will be served during the day.

SUMMARY:
It is a pilot study, conducting on 6 healthy women and aiming at defining new biomarkers related to wheat bran fermentation. For this, a breakfast, containing 5 biscuits enriched in 13-C wheat bran (which grown under 13-CO2 enriched atmosphere) is given to the subjects, then a following will be realized on 24h with breath, urine, fecal and blood samples. Analysis will be performed on these samples in order to determine potential biomarkers of fibers consumption to evaluate the metabolic effects of this consumption and to refine the relevance of nutritional recommendation regarding fibers for healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject able to understand the information given to him and having signed the informed consent form.
* subject having had a medical examination during the selection visit
* Healthy subject
* Female gender
* Age between 20 and 40 years (limits included)
* No Smoking
* Body mass index between 20 and 25 kg / m2 (limits included).
* fiber consumer ≥ 18 g / day
* Do not present any food allergy, nor food intolerance to the products of the study.
* Having no particular diet (vegetarian, vegan, high protein, etc.)
* Having a stool frequency ranging from 1 to 2 per day over the last 2 months
* Absence of pathology detectable by clinical examination and medical examination that may interfere with the evaluation criteria of the study.
* Sedentary subject or practicing steady regular physical activity during the entire study (maximum 4 hours per week).
* Accepting to submit to the protocol of the study with a day of hospitalization of 24h
* Stable weight in the last 3 months (+/- 5% of total body weight)
* Affiliation to a social security scheme.

Exclusion Criteria:

General criteria

* Subject presenting unstable medical or psychological conditions which, according to the investigator, could lead the subject to be non-compliant or uncooperative during the study or could compromise the safety or participation of the subject under study (according to Articles L.1121-6, L.1121-8, L.1121-9 and L1122-1-2 of the Public Health Code).
* Failure to respect the exclusion period of another study specified in the "National Volunteer File".
* Major subject under guardianship.
* Private subject of his liberty by judicial or administrative decision.
* Subject having exceeded the annual amount of compensation for participation in research protocols.
* Not having a refrigerator and / or freezer (necessary for the conservation of collections of urine and / or stool made at home) Biological criteria
* Total blood cholesterol> 11 mmol / L or blood triglycerides> 3 mmol / L
* Fasting blood glucose> 7 mmol / L
* CRP> 10 mg / L
* Demonstration of a biological abnormality judged by the investigator to be clinically significant
* Transaminases (ASAT and ALAT) and gamma GT greater than 1.5 times the upper limit of normal

Medical and therapeutic criteria:

* History of bariatric surgery
* History of digestive surgery with the exception of appendectomy
* Subject presenting gastrointestinal disorders such as ulcers, diverticula or inflammatory bowel diseases
* Diabetes type 1 or 2.
* Chronic renal failure.
* Chronic liver failure.
* known gastroparesis, gastrectomy, colectomy.
* History of chronic gastrointestinal disease with malabsorption.
* External pancreatic insufficiency.
* Known endocrine pathology that can interfere with carbohydrate metabolism (uncontrolled dysthyroidism, acromegaly, hypercorticism, ...).
* Subject with organic intestinal disease.
* subject who has undergone antibiotic therapy in the 3 months preceding the study may interfere with transit or intestinal microbiota:
* Subject treated with a drug that may interfere with carbohydrate metabolism:
* Corticosteroids.
* anorectics.
* High dose gastric bandages.
* Subject having a concomitant pathology incompatible with the constraints of the protocol or which may interfere with the evaluation of the main criterion.
* PA systolic not between 100 and 140 mmHg and diastolic not between 50 and 90 mmHg
* Dieting or wishing to lose weight
* Pregnant woman or wishing to be pregnant or breastfeeding (interrogation data)
* Alcoholism or abuse or dependence on another proven drug. Consumption of more than 3 alcoholic beverages per day is considered abusive. An alcoholic beverage is 30 mL of spirits, 120 mL of wine or 330 mL of beer
* Donation of blood in the 2 months preceding the selection visit
* Subjects consuming dietary supplements
* Subjects refusing to follow the dietary instructions on the 3 days preceding the test day

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Measurement of the 13-C isotopic enrichment kinetics | 24 hours
  Measurement of the 13-C isotopic enrichment kinetics of plasmatic SCFAs after ingestion of 5 biscuits enriched with the 13C-labeled fiber, on 24h.The concentration and the 13C isotopic enrichment of SCFAs in the plasma will be determined according method and tools described by Ferchaud-Roucher and al, 2006 and Ahmed and el, 2016 at the Analyse center of Mass Spectrometry in Lyon

SECONDARY OUTCOMES:
Measurement of the 13-C isotopic enrichment kinetics in CO2 and CH4 from exhaled gases during 24h after fibers ingestion. | 24 hours
  Gases will be taken thanks to the EasySamplerTM Breath Test Kit. The measurements will be done by gas chromatography thanks to a gas analyzer.
Measurement of H2 kinetics in the exhaled breath during 24h. | 24 hours
  H2 will be taken thanks to the EasySamplerTM Breath Test Kit. The measurements will be done by gas chromatography thanks to a gas analyzer.
Measurement of the 13-C isotopic enrichment kinetics of SCFAs in urines after ingestion of 5 biscuits enriched with the 13C-labeled fiber, on 24h. | 24 hours
  The concentration and the 13C isotopic enrichment of SCFAs in the urine will be determined according method and tools described by Ferchaud-Roucher and al, 2006 and Ahmed and el, 2016 at the Analyse center of Mass Spectrometry in Lyon
Measurement of the 13-C isotopic enrichment kinetics of SCFAs in feces after ingestion of 5 biscuits enriched with the 13C-labeled fiber, on 48h or 72h. | Hour 72
  The concentration and the 13C isotopic enrichment of SCFAs in the urine will be determined according method and tools described by Ferchaud-Roucher and al, 2006 and Ahmed and el, 2016 at the Analyse center of Mass Spectrometry in Lyon
The appearance kinetic of 13C glucose in the plasma | 24 hours
  Plasma samples will be prepared and analysed by coupling gas chromatography-combustion-isotopic mass spectrometry according to the method used at the CRNH Rhône-Alpes (Sauvinet et al., 2009)
The platelets aggregation as cardimetabolic risk marker in the plasma | Day -30
  An immuno-enzymatic dosage of platelet thromboxan B2, after the chylomicrons (CM) incubation with platelets, will be done. The measurement of platelet aggregation by aggregometry will be done after the CM and collagen stimulated platelet incubation.
Sphingolipid molecular species concentrations in plasma and TGRL | Day 0
  Isolation of plasma and triglyceride-rich lipoproteins (TGRL) fractions by ultracentrifugation and measurement by liquid chromatography coupled to tandem mass spectrometry (LC-MS/MS)
Fatty acids in lipid classes (triglycerides, phospholipids, cholesteryl esters) of plasma and TGRL | Day 0
  Determination of molar percentages of fatty acids in lipid classes (triglycerides, phospholipids, cholesteryl esters) of plasma and TGRL, following analysis by gas chromatography.
apolipoprotein B48 concentrations in plasma and TGRL | Day 0
  apolipoprotein B48 concentrations in plasma and TGRLby ELISA technique
TGRL particle sizes | Day 0
  TGRL particle sizes by laser granulometry
Intensity of gastro-intestinal symptoms thanks to an analogue visual scale (AVS) | 24 hours
  This AVS allows the measurement of 8 gastro-intestinal symptoms intensity, often described after fibers consumption on a 100 mm scale.
Stool consistency | one week (at each stool)
  Stool consistency by Bristol Stool Chart (type1-7)
Stool frequency | one week
  By questionnaire
Gastro intestinal symptoms | one week
  By questionnaires and visual analogue scale (VAS) score (on a 90mm horizontal line; from no symptom (minimal) to serious symptom (maximum).
measurement of plasmatic PUFA concentration | 24 hours
  Plasma samples will be prepared and analysed by gas-liquid chromatography-
Metagnomic of gut microbiota | one week (at each stool)
  Stool samples will be prepared and analysed by 16SrDBA ilimina sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, MD, Study Director — Centre de Recherche en Nutrition Humaine Rhône-Alpes
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meiller L, Sauvinet V, Breyton AE, Ranaivo H, Machon C, Mialon A, Meynier A, Bischoff SC, Walter J, Neyrinck AM, Laville M, Delzenne NM, Vinoy S, Nazare JA. Metabolic signature of 13C-labeled wheat bran consumption related to gut fermentation in humans: a pilot study. Eur J Nutr. 2023 Sep;62(6):2633-2648. doi: 10.1007/s00394-023-03161-5. Epub 2023 May 24. PMID 37222787
- See also: Related Info — https://www.crnh-rhone-alpes.fr/